CLINICAL TRIAL: NCT05377593
Title: Evaluation of Using Patient Specific Zirconium Dioxide Implant Versus Patient Specific Titanium Implant in Treatment of Chronic Condylar Dislocation. A Randomized Clinical Trial
Brief Title: Evaluation of Using Patient Specific Zirconium Dioxide Implant Versus Patient Specific Titanium Implant in Treatment of Chronic Condylar Dislocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Adham Zakaria, Teaching Assistant at Oral and Maxillofacial Sugery department, Faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMFS 3-3-4
Record Dates: First submitted 2022-05-10; First posted 2022-05-17 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Recurrent Dislocation of Temporomandibular Joint (Disorder)

STUDY DESIGN:
Intervention Model Description: A Randomized Clinical Trial A Trial will be carried out in hospital of Oral and Maxillofacial Surgery department- Faculty of dentistry Cairo University.
  Equal Randomization: Participants receiving treatment. Positive Controlled: Both groups receiving treatment. Parallel group study: each group of patients receives single treatment simultaneously.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eminoplasty with patient specific Titanium onlay implant (Active Comparator)
  Interventions: Device: eminoplasty with patient specific Zirconium dioxide onlay implant
- eminoplasty with patient specific zirconium dioxide onlay implant (Active Comparator)
  Interventions: Device: eminoplasty with patient specific Zirconium dioxide onlay implant

INTERVENTIONS:
Device: eminoplasty with patient specific Zirconium dioxide onlay implant — Eminoplasties will be done for patient with chronic condylar dislocation using patient specific zirconium dioxide implants

SUMMARY:
Alternate hypothesis that treatment of Tempromandibular joint dislocation with Zirconium Dioxide eminoplasty will be more efficient than using titanium onlays in terms of decreasing maximum inter incisal distance and providing better soft tissue response and post-operative patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient with recurrent dislocation with maximum inter incisal opening over 55mm
* Long-standing dislocation of the TMJ involving both fixation for more than 3 weeks and the failure of manual reduction
* Failure of conservative strategies such as orientation to self-limit jaw movement and the use of a chin-cap or bandage
* Both sexes
* Age between 18 and 48 years.
* Highly motivated patients.

Exclusion Criteria:

* Post-menopausal females with osteoporosis
* Patient with uncontrolled systemic disease
* pregnancy
* psychological disorders, drug or alcohol dependency
* Known allergies or sensitivities to dental materials, including Zirconia, Titanium or general anesthetic agents
* Inability to return for follow up visits.
* Refusal of participation from the patient

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Difference in Maximal inter incisal distance between pre-operative and post-operative (mm) | 6 months
  using a caliper the difference between preoperative and postoperative Maximal interincisal opening is recorded (mm)

SECONDARY OUTCOMES:
Patient's Pain | 6 months
  in terms of visual analogue scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Kadry Nasr, Doctorate, Study Director — Lecturer at Oral and Maxillofacial Surgery department, Faculty of dentistry, Cairo University
Locations (1):
- Adham Zakaria, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided